CLINICAL TRIAL: NCT06270680
Title: Efficacy of Carotenoids on Blood Biomarkers Following A Collision Sport Athletes
Brief Title: Carotenoids for Collision Athletes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: MacuHealth (Industry); Orlando Regional Medical Center (Other)
Responsible Party: Principal Investigator, Semyon M. Slobounov, Ph.D., Professor of Kinesiology, Penn State University
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00023019
Record Dates: First submitted 2024-02-03; First posted 2024-02-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Head Injury; Carotenoids
Keywords: Carotenoids; Brain injury; Head impacts; Vision
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplement Group (Experimental): The group receiving the carotenoid supplement.
  Interventions: Drug: Vision Edge Pro
- Placebo Group (Placebo Comparator): The group receiving the placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vision Edge Pro — Each dose will consist of one supplement capsule containing 10 mg lutein, 2 mg zeaxanthin, 10 mg mesozeaxanthin, 50mg EPA, 250mg DHA. Capsules are to be taken orally, once daily with a meal. Duration of supplementation will last approximately 2 - 5 months, depending on the length of the athletic seasons for the sports recruited.
  Other Names: Carotenoid supplement
  Arms: Supplement Group
Other: Placebo — A sunflower oil placebo containing 380 mg of sunflower oil
  Arms: Placebo Group

SUMMARY:
This is a supplement study being conducted to find out if collision sport athletes who are exposed to repetitive head impacts while supplementing with carotenoids will have decreased pro-inflammatory blood biomarkers, increases in macular pigment optical density, improved contrast sensitivity, greater retinal nerve fiber thickness, and better overall visual quality of life scores compared to collision athletes taking a placebo.

DETAILED DESCRIPTION:
Originally adapted to augment macular pigment for anti-inflammatory, antioxidative, blue light, and visual performance purposes, supplementation with carotenoids has been tested in animal models for protective effects against traumatic brain injury (TBI). Results have been promising, as mice provided with the three main carotenoids (Lutein, Meso-Zeaxanthin, and Zeaxanthin) following TBI displayed reduced levels of pro-inflammatory markers (IL-1β, IL-6, and GFAP) and increased levels of GAP43, NCAM, and BDNF, signaling activation of anti-oxidant systems.

Due to inflammation of the visual system following trauma, immune responses in the eye are for both reparative and protective purposes. However, cytokines released by immune cells compromise visual acuity by means of inflammation and fibrosis (scarring). As such, inflammation to the visual system (including visual processing structures in the brain) carries the danger of visual impairment. Research examining chronic inflammatory responses in the optic tract and subsequent visual dysfunction found mTBI in rodent models to increase GFAP, tumor necrosis factor (TNF), and degeneration of axons up to 3.5 months post-injury. As such, inflammation of the visual system is a measurable phenomenon in rodent models, conveying the need for human subjects research. The nutrients found in the proposed test supplement, lutein, zeaxanthin, meso-zeaxanthin, along with the omega-3 fatty acids DHA and EPA, are deposited in the brain regions that are often found to be affected by a collision-related head injury. Thus, an exploratory study of this topic is proposed, utilizing the three main carotenoids in the form of a MacuHealth supplement.

Optical Coherence Tomography has become a critical clinical tool when discovering and diagnosing disease and neurological disorders of the eyes. It works to map the retina in order to give ophthalmologists precise measurements of the tissues which make up this important part of human anatomy and helps medical experts to diagnosis diseases of the eye such as Glaucoma and Macular Degeneration. In terms of retinal nerve fiber layer thickness (RNFL), a study found Olympic boxers to have thinner RNFL compared to controls. Another study found RNFL thickness as a significant predictor of athlete vs control status, with 4.8-um of thinning seen on average in athletes (boxing, football) when compared to controls.

Although vision disorders are so common, VQOL - to our knowledge - is not specifically addressed following exposure to repetitive head impacts (RHI), concussion, or during return-to-play protocol. In sports such as football, hockey, and boxing where participants are exposed to RHI, participation while experiencing decreased VQOL or visual functionality could prove costly to the health of those athletes. Poor visual acuity and photophobia following concussion have been cited as indicators of poor VQOL. As such, use of the VFQ-25 and the 10-Item Supplement may be important additions to current clinical practice when evaluating the baseline health status of athletes, and following the completion of a collision-sport season.

ELIGIBILITY:
Inclusion Criteria:

* Collision sport athletes:

  1. Penn State student ages 18 and over
  2. Any gender
  3. Participating in club, or intramural collision-sports and is willing to participate in this study (examples: hockey, lacrosse, soccer, wrestling, rugby, boxing, basketball, cheer).

Exclusion Criteria:

* For all subjects:

  1. Subjects with concurrent injury that would impair their ability to perform the assigned procedures will be excluded.
  2. Under 18 years of age.
  3. Not a Penn State Student
  4. Not participating in a collision sport.
  5. Diagnosis of a learning disability impacting their capacity to consent.
  6. History of ocular or neurological disease (glaucoma, macular degeneration, MS, Parkinson's)
  7. Concussion diagnosis within the last calendar year.
* However, if a subject sustains a concussion during the course of the study, they may remain as an active participant if they wish to do so.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Blood and saliva biomarkers via venous blood draw and spitting into sterile cup. | Up to 16 weeks
  1. To explore the effect of Lutein, Meso-Zeaxanthin, and Zeaxanthin supplementation on blood and saliva biomarkers following a single competitive season of collegiate collision sport. Specific markers will include GFAP, NF-L, UCH-L1, SBDP, Tau, S100B, BDNF, IL-1B, IL-6.
Visual Performance: Speed of visual processing | Up to 16 weeks
  2. To assess the visual performance parameter of speed of visual processing, measured in hertz (Hz). Measured using a densitometer.
Visual Performance: Contrast Sensitivity | Up to 16 weeks
  3. To assess visual performance parameter of contrast sensitivity, measured by the percentage threshold of contrast reached using M&S Technologies Smart System Software.
Skin carotenoid concentration | Up to 16 weeks
  4. To measure skin carotenoid concentration to ensure compliance and bioavailability of the test supplement.
Retinal Nerve Fiber Layer Thickness | Up to 16 weeks
  5. Utilize Optical Coherence Tomography to examine changes in retinal nerve fiber layer thickness (RNFL) following exposure to repetitive head impacts during a single competitive season of collision sports.
Macular Pigment Optical Density | Up to 16 weeks
  6. To explore the effect of Lutein, Meso-Zeaxanthin, and Zeaxanthin supplementation on macular pigment optical density (MPOD) following supplementation over the course of a collegiate season. This is the measurement of blue light reduction by macular pigment, related to the amount of macular pigment carotenoids in an individual's body. Measured using densitometer.
Visual Quality of Life Scores | Up to 16 weeks
  7. To explore the effect of Lutein, Meso-Zeaxanthin, and Zeaxanthin supplementation on self-reported measures of visual quality of life (VQOL) using the National Eye Institute Visual Functioning Questionnaire-25 (VFQ-25). Scale title: The National Eye Institute 25-Item Viual Function Questionnaire; minimum value of 0, maximum value of 100; higher score means a better outcome.
Visual Quality of Life Scores | Up to 16 weeks
  8. To explore the effect of Lutein, Meso-Zeaxanthin, and Zeaxanthin supplementation on self-reported measures of visual quality of life (VQOL) using the 10-Item Neuro-Ophthalmic Supplement (10-Item Supplement). Scale title: Ten Item Neuro-Ophthalmic Supplement; minimum value of 0, maximum value of 100; higher score means a better outcome.

SECONDARY OUTCOMES:
Demographic information | Up to 16 weeks
  Secondary endpoints that will be measured are headache or migraine history, history of learning disability, dyslexia, ADD/ADHD, self- and family-history of psychiatric disorder. Recorded with yes or no answers.
Demographic information | Up to 16 weeks
  Secondary endpoints that will be measured are duration of sport participation each week, measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Semyon Slobounov, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stringham JM, Hammond BR. Macular pigment and visual performance under glare conditions. Optom Vis Sci. 2008 Feb;85(2):82-8. doi: 10.1097/OPX.0b013e318162266e. PMID 18296924
- [Background] Stringham JM, Stringham NT, O'Brien KJ. Macular Carotenoid Supplementation Improves Visual Performance, Sleep Quality, and Adverse Physical Symptoms in Those with High Screen Time Exposure. Foods. 2017 Jun 29;6(7):47. doi: 10.3390/foods6070047. PMID 28661438
- [Background] Stringham JM, Johnson EJ, Hammond BR. Lutein across the Lifespan: From Childhood Cognitive Performance to the Aging Eye and Brain. Curr Dev Nutr. 2019 Jun 4;3(7):nzz066. doi: 10.1093/cdn/nzz066. eCollection 2019 Jul. PMID 31321376
- [Background] Gunal MY, Sakul AA, Caglayan AB, Erten F, Kursun OED, Kilic E, Sahin K. Protective Effect of Lutein/Zeaxanthin Isomers in Traumatic Brain Injury in Mice. Neurotox Res. 2021 Oct;39(5):1543-1550. doi: 10.1007/s12640-021-00385-3. Epub 2021 Jun 15. PMID 34129176
- [Background] Stepp MA, Menko AS. Immune responses to injury and their links to eye disease. Transl Res. 2021 Oct;236:52-71. doi: 10.1016/j.trsl.2021.05.005. Epub 2021 May 27. PMID 34051364
- [Background] Chen JJ, Bhatti MT. Papilledema. Int Ophthalmol Clin. 2019 Summer;59(3):3-22. doi: 10.1097/IIO.0000000000000274. No abstract available. PMID 31233413
- [Background] Vishwanathan R, Neuringer M, Snodderly DM, Schalch W, Johnson EJ. Macular lutein and zeaxanthin are related to brain lutein and zeaxanthin in primates. Nutr Neurosci. 2013 Jan;16(1):21-9. doi: 10.1179/1476830512Y.0000000024. Epub 2012 Jul 9. PMID 22780947
- [Background] Strong J. Retinal OCT Imaging - Ophthalmic Photographers' Society. Published 2011. Accessed January 5, 2023. https://www.opsweb.org/page/RetinalOCT
- [Background] Childs C, Barker LA, Gage AM, Loosemore M. Investigating possible retinal biomarkers of head trauma in Olympic boxers using optical coherence tomography. Eye Brain. 2018 Dec 14;10:101-110. doi: 10.2147/EB.S183042. eCollection 2018. PMID 30588143
- [Background] Leong D, Morettin C, Messner LV, Steinmetz RJ, Pang Y, Galetta SL, Balcer LJ. Visual Structure and Function in Collision Sport Athletes. J Neuroophthalmol. 2018 Sep;38(3):285-291. doi: 10.1097/WNO.0000000000000572. PMID 28885451
- [Background] Armstrong RA. Visual problems associated with traumatic brain injury. Clin Exp Optom. 2018 Nov;101(6):716-726. doi: 10.1111/cxo.12670. Epub 2018 Feb 28. PMID 29488253